CLINICAL TRIAL: NCT06382883
Title: The Impact of Individually Tailored Lifestyle and Physical Activity Intervention on Obstructive Sleep Apnea in Overweight, CPAP-treated Patients in Finland: A Randomized Controlled Trial
Brief Title: Lifestyle and Physical Activity as Part Of Obstructive Sleep Apnea Treatment
Acronym: ELO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Filha ry (Other)
Collaborators: University of Jyvaskyla (Other); Organisation for Respiratory Health in Finland (Unknown); Central Finland Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FINELO2024
Record Dates: First submitted 2024-04-03; First posted 2024-04-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; physical activity; sedentary behavior; behavioral change
MeSH Terms: conditions — Sleep Apnea, Obstructive; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEMC-protocol (Experimental): Assigned participants will receive CPAP-therapy and one year individually tailored lifestyle intervention at the Sports Medicine Outpatient Clinic of The Wellbeing Services County of Central Finland (SEMC).
  Interventions: Behavioral: Individually tailored lifestyle and physical activity intervention
- SEMC-protocol + EBS intervention (Experimental): Assigned participants will receive CPAP-therapy, SEMC-protocol as described above and enhanced behavioral support -intervention (EBS). The EBS-intervention will apply a patient-centered self-regulatory approach to support (motivation for) changes in behavior (CPAP-use, physical activity (PA), and sedentary behavior (SB)).
  Interventions: Behavioral: Individually tailored lifestyle and physical activity intervention combined with enhanced behavioral support -intervention (EBS)
- Control group (No Intervention): Assigned participants will receive CPAP-therapy, receive written information on healthy lifestyle but will not receive any extra support.

INTERVENTIONS:
Behavioral: Individually tailored lifestyle and physical activity intervention — Focus of the SEMC-protocol is on increasing PA gradually towards the national recommendations. Emphasis of counseling is on incidental exercise, endurance, and strength training. Techniques of motivational interviewing are utilized.
  Baseline; MD+PT counseling, medical clearance, mapping lifestyle & life situation, goal setting, measurements, questionnaires, feedback. weeks 1-6: guided group resistance training 1hr, 1x/week. 5-10-minute warm-up, 9 exercises with weight stack equipment on large muscle groups. 2-3 sets, 12-15 repetitions. Modified individually, e.g. according to musculoskeletal problems. Emphasis on learning the basics and safety aspects. After 6 weeks unsupervised training. 3-month: MD counseling and questionnaires. 6-month: MD+PT counseling, assessing safety of PA, measurements, questionnaires, feedback. 12-month: MD+PT counseling (feedback, ensuring continuity of lifestyle changes; redirecting to municipality/NGO activities), measurements, questionnaires, feedback
  Other Names: SEMC-protocol
  Arms: SEMC-protocol
Behavioral: Individually tailored lifestyle and physical activity intervention combined with enhanced behavioral support -intervention (EBS) — In addition to the SEMC-protocol, the participants will be contacted 3 times during the first 3 months (live / online as preferred). Themes:
  Session 1: Motivation and illness perceptions. Exploring CPAP use, PA, and SB. Session 2: Self-regulation (feedback, goal setting, self-monitoring, action planning, problem solving), activating social support, prompts/cues, and preparatory behaviors. (Included BCTs from Michie et al 2013 taxonomy: 3.2, 12.2, 8.3,) Session 3: Assessing progress and agenda setting, self-regulation, maintenance of PA.
  Measurements and questionnaires as with SEMC-protocol.
  Other Names: SEMC-protocol + EBS intervention
  Arms: SEMC-protocol + EBS intervention

SUMMARY:
The goal of this clinical trial is to investigate the effects of an individually tailored lifestyle intervention on symptoms and severity of obstructive sleep apnea (OSA), physical activity (PA) levels and sedentary behavior (SB), as well as health and wellbeing in overweight participants with moderate to severe OSA treated with CPAP. Emphasis of the individually tailored SEMC-intervention (protocol of the Sports Medicine Outpatient Clinic of The Wellbeing Services County of Central Finland) is on increasing the amount of total physical activity.

The main questions the trial aims to answer are:

* Can individually tailored lifestyle intervention, in combination with CPAP therapy, alleviate the severity or symptoms of OSA in overweight participants with moderate to severe OSA?
* Does the addition of an individually tailored lifestyle intervention to CPAP therapy improve the quality of life, increase physical functioning, change body composition, and increase physical activity levels or decrease sedentary behavior of participants diagnosed with moderate to severe OSA?
* Can enhanced behavioral support (EBS), when integrated with lifestyle intervention and CPAP therapy, lead to more substantial and enduring changes in participants' levels of physical activity or sedentary behavior?

Participants will be randomized to either SEMC-intervention group, combination of SEMC-intervention and EBS, or to a control group.

In this study, it is hypothesized that participants receiving SEMC-intervention in combination with CPAP therapy will experience greater alleviation of OSA severity and symptoms, improve their quality of life, body composition and physical functioning, as well as increase physical activity levels and decrease their sedentary behavior compared to the control group. In addition, it is hypothesized that participants receiving SEMC-intervention and EBS in combination with CPAP therapy will increase their physical activity levels, and decrease their sedentary behavior to a greater extent, and these changes will be more sustained compared to merely SEMC-intervention or control group.

DETAILED DESCRIPTION:
Approximately 400,000 adults in Finland are diagnosed with obstructive sleep apnea (OSA). The prevalence of OSA has dramatically increased during the past years. It is estimated that substantial number of patients remain undiagnosed. Untreated OSA is associated with multiple chronic diseases causing increased morbidity, mortality, and health care costs in the western countries. Approximately 70% of patients with OSA are overweight, which is the most common risk factor of OSA.

While CPAP therapy often effectively alleviates symptoms of OSA, it usually does not address the underlying issue, as body weight often remains unchanged or even increases with CPAP therapy, especially among young and women. Additionally, CPAP therapy has limited impact on cardiometabolic risk factors, which commonly accumulate in patients with OSA. Exercise, even without significant weight loss, has been shown to positively impact the severity of OSA and its symptoms, as well as several cardiometabolic risk factors. Not to mention the additional benefits of sustained weight reduction.

Previous research has focused on exercise interventions that are similar for all participants. There are only few studies executed in clinical, real-life setting or studies with long-term follow-up periods.

This clinical trial aims to investigate whether an individually tailored lifestyle intervention (SEMC-protocol) aimed at increasing physical activity levels will affect the severity or symptoms of OSA, participants' quality of life, their cardiometabolic risk factors, anthropometry, functional capacity, or induce lasting behavioral changes (physical activity and sedentary behavior). This trial also investigates whether enhanced behavioral support (EBS) will lead to more substantial and enduring changes in participants' levels of physical activity and sedentary behavior.

The participants (n=300) will be recruited at the respiratory outpatient clinic of central Hospital Nova in Jyväskylä, Finland. Information of the clinical trial will be provided to potential participants when starting CPAP therapy according to standard treatment. The candidates will sign a written consent for a phone call from a researcher providing more information on the study. After the phone call, they will decide whether to sign the final informed consent to participate in the study.

Participants are randomly allocated to either SEMC-intervention group, combination of SEMC-intervention and EBS-intervention, or to a control group. Comparisons between the groups are made at 3, 6 and 12months after baseline. Additionally, long-term assessments of the participants' health status are assessed from registry data and via questionnaires at 2-, 3-, and five-year follow-up studies.

Ethical approval for this study was obtained from the Ethics Committee of The Wellbeing Services County of Central Finland in August 2023.

In the power calculations and sample size determination, based on previous literature it was assumed that the change in apnea-hypopnea-index (AHI) for the intervention group is at least 10/h ± 10, and for the controls it is 5 ± 10 /h. Thus, the sample size should be at least 126 participants (63 in the intervention group and 63 in the control group) when the type I error probability is 0.05 and the type II error probability is 0.2. With this sample size, the power is 0.8 (80%). Assuming a dropout rate of at least 10% for the study, 100 participants will be enrolled in both the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* A physician-diagnosed, moderate to severe obstructive sleep apnea
* BMI > 25
* Age 18- to 70-years
* No previous CPAP-treatment

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD) or other severe conditions affecting nighttime oxygenation (mild asthma is acceptable), Obesity Hypoventilation Syndrome without sleep apnea.
* Aggressive cancer or any other condition requiring intense treatments.
* Weight-loss medication initiated less than 3 months before recruiting
* Conditions severely impairing daily functioning (e.g., serious mental health issues, narcolepsy, severe comorbidities, profound fibromyalgia, musculoskeletal problems significantly limiting mobility and accordingly, participation in the intervention)
* Conditions and diseases influencing the participant's ability to make independent decisions
* Participants under 18 years of age
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in apnea-hypopnea-index (AHI) | Assessed at pre-intervention, and 12 months.
  Measured with sleep polygraphy (SomnoMedics), analyzed by an experienced professional according to current guidelines.

SECONDARY OUTCOMES:
Change on sleep apnea symptoms | Assessed at base line, 3 months, 6 months, and 12 months.
  Symptoms typically associated with OSA are measured by a questionnaire on the amount and severity of symptoms experienced during the last week prior filling the questionnaire, on a scale from 0 to 10, 0 being "not at all" and 10 "all the time". The symptoms asked are according to Finnish OSA diagnosis and treatment guidelines.
Change in the mean daily total light physical activity time | Time Frame: Assessed by questionnaire at base line, 3 months, 6 months, and 12 months (and 2, 3 and 5 years) and by SENS Motion® Activity Measurement System at base line and 6 months.
  Measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF) and SENS Motion® Activity Measurement System (assessed with 7-day recordings).
Change in the mean daily total moderate to vigorous (MVPA) physical activity time | Time Frame: Assessed by questionnaire at base line, 3 months, 6 months, and 12 months (and 2, 3 and 5 years) and by SENS Motion® Activity Measurement System at base line and 6 months.
  Measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF) and SENS Motion® Activity Measurement System (assessed with 7-day recordings).
Change in the mean daily total sedentary time | Time Frame: Assessed by questionnaire at base line, 3 months, 6 months, and 12 months (and 2, 3 and 5 years) and by SENS Motion® Activity Measurement System at base line and 6 months.
  Measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF) and SENS Motion® Activity Measurement System (assessed with 7-day recordings). The IPAQ-SF is a concise self-assessment tool comprising 7 items designed to evaluate the duration and intensity of physical activity (PA) and sedentary behavior within individuals' daily routines over the preceding 7 days.
Change in 6-minute walk distance (6MWD) in meters | Assessed at base line, 6 months, 12 months
  Measured by 6-minute-walk test (6MWT), according to the guidelines of the American Thoracic Society (ATS).
Change in hand grip strength in kilograms | Assessed at base line, 6 months, 12 months
  Measured by Saehan SH5001 hand dynamometer
Change in waist circumference in centimeters | Assessed at base line, 6 months, 12 months
  Waist circumference in centimeters.
Change in body weight in kilograms | Assessed at base line, 6 months, 12 months
  Weight in kilograms, measured by Bioelectrical Impedance Analysis (InBody770 body composition analyzer, Biospace Co. Ltd, Seoul, South Korea)
Change in visceral fat area (VFA) in square centimeters | Assessed at base line, 6 months, 12 months
  Visceral fat area in square centimeters. Measured by Bioelectrical Impedance Analysis (InBody770 body composition analyzer, Biospace Co. Ltd, Seoul, South Korea)
Change in muscle mass in kilograms | Assessed at base line, 6 months, 12 months
  Muscle mass in kilograms. Measured by Bioelectrical Impedance Analysis (InBody770 body composition analyzer, Biospace Co. Ltd, Seoul, South Korea)
Change in Quality of Life RAND 36-Item Health Survey | Assessed at base line, 3 months, 6 months, and 12 months (and 2, 3 and 5 years)
  Measured by RAND-36 questionnaire. The RAND 36 questionnaire is a self-report instrument comprising 36 items designed to evaluate eight dimensions of general health status over the preceding four weeks. Responses to the questionnaire are quantified using a numeric scale ranging from 0 (minimum score) to 100 (maximum score), with higher scores indicating better health outcomes. Subsequently, these scores are expressed as a percentage of the total possible score. Items within each dimension are averaged to derive the respective scale scores. Any unanswered items (missing data) are disregarded in the computation of scale scores. Consequently, the scale scores reflect the average of all answered items within the respective dimension.

CONTACTS AND LOCATIONS:
Overall Officials: Tuula Vasankari, Principal Investigator — Filha ry (Finnish Lung Health Association)
Locations (1):
- Central Finland Hospital District, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: No